CLINICAL TRIAL: NCT02974699
Title: Role of Gastrointestinal Microbes on Digestion of Resistant Starch and Tryptophan Availability to Humans
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Wayne State University (Other)
Responsible Party: Principal Investigator, Paul Burghardt, Assistant Professor, Wayne State University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 110116M1F
Record Dates: First submitted 2016-11-21; First posted 2016-11-28 (Estimated); Last update posted 2017-05-04 (Actual); Status verified 2017-05

CONDITIONS: Type II Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Potato Starch (Bob's Red Mill) (Experimental): Daily dietary supplementation with Potato Starch (48g total/day) suspended in water. 24g will be consumed 2 times per day.
  Interventions: Dietary Supplement: Potato Starch (Bob's Red Mill)
- Resource ThickenUp Pregelatinized Starch (Placebo Comparator): Daily dietary supplementation with Pregelatinized Starch (48g total/day) suspended in water. 24g will be consumed 2 times per day.
  Interventions: Dietary Supplement: Pregelatinized Starch (Resource ThickenUp)

INTERVENTIONS:
Dietary Supplement: Potato Starch (Bob's Red Mill) — Subjects will be assigned to Potato Starch (active) following assessment of their gut microbiome.
  Arms: Potato Starch (Bob's Red Mill)
Dietary Supplement: Pregelatinized Starch (Resource ThickenUp) — Subjects will be assigned to Pregelatinized Starch (placebo) following assessment of their gut microbiome.
  Arms: Resource ThickenUp Pregelatinized Starch

SUMMARY:
There is currently a critical gap in knowledge of how intestinal bacterial communities alter metabolic substrates available to the host thereby influencing central and enteric nervous system (CNS/ENS) neurotransmitter levels involved in regulating carbohydrate consumption in humans. Understanding these relationships is essential for developing strategies to improve blood glucose control and to reduce the risk of transitioning from prediabetes to type-2 diabetes (T2D). The investigators' long-term goal is to determine the biological underpinnings of behaviors that impact food intake and blood glucose control that contribute to the development of T2D. The objective of this proposal, which is an essential next step in attaining the investigators' long-term goals, is to determine how bacterial populations in the digestive system impact circulating tryptophan (TRP) and large neutral amino acid (LNAA) levels that regulate production of monoamine 5-hydroxytryptamine (5-HT, serotonin) in the ENS and in gastrointestinal system and the brain. The central hypothesis is that a reduced ratio of TRP producing (TRPp) to TRP consuming (TRPc) bacteria (decreased TRPp:TRPc ratio) in the gut will decrease TRP availability following a carbohydrate meal lowering the plasma TRP:LNAA ratio and resulting in less TRP for ENS/CNS production of 5HT. Further, dietary interventions that promote TRPp bacterial abundance within the gut will increase TRP availability to the host. The investigators will test the central hypothesis and, thereby, accomplish the overall objective for this project by pursuing the following specific aims: 1) Assess impact of divergent microbiota on plasma TRP:LNAA ratio in response to acute carbohydrate consumption, and 2) Assess the impact of dietary supplementation with resistant starch (RS) on gut microbiota and circulating TRP:LNAA ratio. During Aim 1, stool samples will be collected from healthy participants. Participants will be stratified based on gut TRPp:TRPc ratio and the response to an acute meal will be assessed by determining plasma TRP:LNAA ratios. During Aim 2 the capacity for 4-weeks of pre-biotic RS (Potato Starch) supplementation to increase the TRPp:TRPc bacterial ratio in the gut will be determined from stool samples. Additionally, plasma TRP:LNAA ratio following acute carbohydrate consumption before and after supplementation will be determined. The scientific contribution will be to determine the impact of RS on TRPp and TRPc bacteria abundance in the gut, and how bacterial populations impact circulating TRP:LNAA levels, that can impact ENS and CNS 5HT production in humans. This contribution will be significant because it will have direct translational implications for human diseases with altered 5HT signaling.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female
2. Age 18 - 65 years old
3. Non-Obese (BMI ≤ 30 kg/m2 and >17 kg/m2 )

Exclusion Criteria:

1. Urine toxicology positive,
2. Pregnant (female)
3. Alcohol intake 48 hours prior to studies,
4. Evidence of inherited disorders of lipid metabolism,
5. History of Cancer within the last 5 years,
6. Human immunodeficiency virus (HIV) antibody positive,
7. Patients with solid organ transplants,
8. Unstable angina or NY heart association class II failure or above,
9. Gastrointestinal disease specifically GI motility disorders,
10. Unstable neuropsychiatric disease including major depression/anxiety, eating disorder such as bulimia or anorexia,
11. End stage renal or hepatic disease,
12. Autoimmune disorders (e.g. SLE),
13. Prior bariatric surgery,
14. A history or current alcohol/substance abuse or nicotine containing products or illicit drugs of abuse during the preceding 6 months,
15. Treatment within one month with sedative hypnotic medications (benzodiazepines, barbiturates), or over the counter sleeping aids
16. Women: any selective estrogen receptor modulator or aromatase inhibitor Men:

    androgen ablation/deprivation hormonal therapies
17. Any medical condition, which in the opinion of the investigator would make the patient unsuitable for recruitment, or could interfere with the patient participating in or completing the protocol
18. Any previous adverse events or allergic reactions to acetaminophen
19. Unwilling or unable to consent for the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2017-01; Primary Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Plasma Amino Acid Levels | Baseline
Plasma Amino Acid Levels | Following 4 weeks of supplementation

SECONDARY OUTCOMES:
Change in Plasma Amino Acid Levels | Baseline vs. 4-weeks
  Difference in plasma amino acid levels between baseline and following 4-weeks of supplementation

CONTACTS AND LOCATIONS:
Locations (1):
- Wayne State University, Detroit, Michigan, United States